CLINICAL TRIAL: NCT06335797
Title: Optimization of Postoperative Bowel Habits Following Pelvic Reconstructive Surgery: a Randomized Controlled Trial
Brief Title: Optimization of Postoperative Bowel Habits
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00110733
Record Dates: First submitted 2024-03-22; First posted 2024-03-28 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-03

CONDITIONS: Constipation
Keywords: Bowel Habits; Pelvic Surgery; Laxatives
MeSH Terms: conditions — Constipation | interventions — Sennosides

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- SENNA (Experimental): Group A participants will be prescribed oral senna (Senokot; Atlantis Consumer Healthcare Inc., Bridgewater, NJ) 8.6mg tablets and be instructed to start with two tablets on the morning of Post Operative Day (POD)#1. Participant will continue taking two tablets on the daily. If no bowel movement on the morning of POD#3 participant may take 2 tablets in the morning and another 2 tablets that evening. The same can be replicated on POD#4. If no bowel movement on the morning of POD#5 participant may take magnesium hydroxide (Phillips' Milk of Magnesia; Bayer AG, Leverkusen, Germany) 30 mL by mouth and need to call the urology clinic for further instruction.
  Interventions: Dietary Supplement: Senna Tab
- DULCOLAX (Experimental): Group B participants will be prescribed bisacodyl rectal (Dulcolax Suppository; Sanofi S.A., Paris, France) 1 suppository to be placed rectally on the morning of Post Operative Day (POD)#1. Participant will continue placing a nightly rectal suppository until their first bowel movement. If no bowel movement by the morning of POD#5 participant may take magnesium hydroxide (Phillips' Milk of Magnesia; Bayer AG, Leverkusen, Germany) 30 mL by mouth and need to call the clinic for further instruction.
  Interventions: Dietary Supplement: Dulcolax Suppositories

INTERVENTIONS:
Dietary Supplement: Senna Tab — Senna 8.6mg two tablets per day post operative day 1 and and if needed, then continue on the same dose regiment until post operative day 5.
  Other Names: Senokot
  Arms: SENNA
Dietary Supplement: Dulcolax Suppositories — Dulcolax 1 suppository to be placed rectally on the evening of post operative day 1 and if needed, then continue using the same dose regiment until the post operative day 5.
  Other Names: Bisacodyl Suppositories
  Arms: DULCOLAX

SUMMARY:
Project is a trial, in which women undergoing vaginal surgery for pelvic organ prolapse will be randomized 1:1 to a postoperative bowel regimen of either oral senna or rectal bisacodyl suppository.

DETAILED DESCRIPTION:
Delayed return to bowel function following vaginal surgery for pelvic organ prolapse has been deemed to be highly distressing for patients, and is ranked as one of the most common reasons for emergency department visits and telephone calls in the immediate post-operative period.

Despite the prevalence of constipation and significant effect on quality of life, few studies have examined an evidence-based bowel regimen for postoperative constipation prevention in the Urogynecology population.

As per available medical literature, the onset of action for oral senna occurs within 6-12 hours, while bisacodyl suppository can take effect between 15 and 60 minutes following rectal administration. Proposed trial comparing oral senna to rectal bisacodyl suppositories for the prevention of postoperative constipation in women undergoing vaginal reconstructive surgery for symptomatic prolapse.

ELIGIBILITY:
Inclusion Criteria:

* Women ages 18 and older scheduled to undergo vaginal pelvic organ prolapse repair

Exclusion Criteria:

* Women younger than 18 years old
* Those unable to provide consent
* Preexisting chronic laxative use
* Conditions that could affect bowel function including, inflammatory bowel disease, irritable bowel syndrome, colorectal cancer, rectovaginal fistula; concurrent bowel surgery; intraoperative bowel injury

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — This is a randomized clinical trial in women getting vaginal reconstructive surgery for correction of bothersome pelvic organ prolapse.
Enrollment: 88 (Estimated)
Dates: Start 2024-10-16 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Time in hours to first bowel movement comparison between the two arms | up to Post Operative Day (POD) 5
  To compare the time to first bowel movement after use of bisacodyl suppositories or oral senna in women undergoing vaginal reconstructive surgery for pelvic organ prolapse. Time in hours will be recorded from the end of the surgical procedure. That is Post Operative Day (POD) 0. First bowel movement will be recorded up to POD5.

SECONDARY OUTCOMES:
Change in Overall Satisfaction (TSQM) Scores | Day 7
  Patients will complete the Treatment Satisfaction Questionnaire for Medicine (TSQM) at 1 week postop. The TSQM is a validated survey assessing patient satisfaction to treatment - It consists of 14 questions, with 7 possible answers for each question, ranging from "extremely agree" to extremely disagree. Higher Scores meaning more satisfaction.
Visual Analog Scale (VAS) Pain Scores | Post Operative Day (POD)1, POD2, POD3, POD4, and POD5
  Patients will be asked to rate their pain with first bowel movement using an 11-point visual analog scale (VAS), in which a score of 0 equates to "no pain" and a score of 10 equates to the "worst pain possible." - VAS ratings of 0 to 4 mm can be considered no pain; 5 to 44 mm, mild pain; 45 to 74 mm, moderate pain; and 75 to 100 mm, severe pain.
Patient Assessment of Constipation Symptom Questionnaire (PAC-SYM) Scores | Baseline and Day 7
  The Patient Assessment of Constipation Symptom Questionnaire is a validated 12-item questionnaire based on the Rome criteria for constipation and is tailored to assess a change in short-term constipation symptoms after an intervention. A score of 0.35 or greater on the Patient Assessment of Constipation Symptom Questionnaire is consistent with constipation, and the changes in scores correlate with clinical changes in constipation symptoms. Items are scored on 5-point Likert scales, with scores ranging from 0 to 4 (0 = 'symptom absent', 1 = 'mild', 2 = 'moderate', 3 = 'severe' and 4 = 'very severe').
Bristol Stool Form Scale (BSFS) Scores | Post Operative Day (POD)1, POD2, POD3, POD4, and POD5
  The Bristol Stool Form Scale (BSFS) is a visual bowel movement rating scale from 1 to 7 that provided a validated measure of gut transit time based on the shape, consistency, and appearance of the bowel movement. The BSFS is an ordinal scale of stool types ranging from the hardest (type 1) to the softest (type 7) that is widely used in practice and clinical research to measure stool form. Types 1 and 2 are considered abnormally hard stools (and in conjunction with other symptoms indicative of constipation).

CONTACTS AND LOCATIONS:
Overall Officials: Candace Parker-Autry, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Caljouw MA, Hogendorf-Burgers ME. GYNOTEL: telephone advice to gynaecological surgical patients after discharge. J Clin Nurs. 2010 Dec;19(23-24):3301-6. doi: 10.1111/j.1365-2702.2010.03395.x. Epub 2010 Oct 14. PMID 20946445
- [Background] Ramaseshan AS, LaSala C, O'Sullivan DM, Steinberg AC. Patient-Initiated Telephone Calls in the Postoperative Period After Female Pelvic Reconstructive Surgery. Female Pelvic Med Reconstr Surg. 2020 Oct;26(10):626-629. doi: 10.1097/SPV.0000000000000636. PMID 30247168
- [Background] Arya LA, Novi JM, Shaunik A, Morgan MA, Bradley CS. Pelvic organ prolapse, constipation, and dietary fiber intake in women: a case-control study. Am J Obstet Gynecol. 2005 May;192(5):1687-91. doi: 10.1016/j.ajog.2004.11.032. PMID 15902178
- [Background] Patel M, Schimpf MO, O'Sullivan DM, LaSala CA. The use of senna with docusate for postoperative constipation after pelvic reconstructive surgery: a randomized, double-blind, placebo-controlled trial. Am J Obstet Gynecol. 2010 May;202(5):479.e1-5. doi: 10.1016/j.ajog.2010.01.003. Epub 2010 Mar 6. PMID 20207340
- [Background] Tarumi Y, Wilson MP, Szafran O, Spooner GR. Randomized, double-blind, placebo-controlled trial of oral docusate in the management of constipation in hospice patients. J Pain Symptom Manage. 2013 Jan;45(1):2-13. doi: 10.1016/j.jpainsymman.2012.02.008. Epub 2012 Aug 11. PMID 22889861